CLINICAL TRIAL: NCT05647837
Title: Value of Cerebrospinal Fluid (CSF) Biomarkers in Patients of Idiopathic Intracranial Hypertension (IIH) as an Indicative of Visual Affection and Treatment Modalities
Brief Title: CSF Biomarkers in Idiopathic Intracranial Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ebrahim Ahmed Yousof Abdelhakeem, principle investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSF biomarkers
Record Dates: First submitted 2022-10-22; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-11

CONDITIONS: Intracranial Hypertension
Keywords: biomarkers
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients wit IIH (Experimental): patient that complains of symptoms of chronic increase intracranial pressure especially visual with absent of organic cause through visual assessment, routine laboratory investigation and brain imaging.
  these patients will undergo lumper puncture to assess CSF opening pressure and Neurofilament Light Chain (NFL) and HYpoxia Induced Factor (HIF) both in CSF and blood.
  Interventions: Diagnostic Test: lumper puncture

INTERVENTIONS:
Diagnostic Test: lumper puncture — lumper puncture

SUMMARY:
Aim of the study is to high lighten the rule of CSF biomarkers in early diagnosis of IIH and in follow up to reach to a definite clinically based decision if this patient will improved on medical treatment or that patient is in need for surgical intervention.

DETAILED DESCRIPTION:
Idiopathic intracranial hypertension (IIH) is a rare disease of increasing incidence recently[1], owing to the rising curve of obesity and weight gain[2,3]. It is a disease of elevated intracranial pressure without known obvious aetiology. The reported incidence of IIH is 1 to 3 cases per 100,000 people of the general population[4]. IIH is diagnosed by exclusion; as patients come with continuous headache repeated vomiting , pulsatile tinnitus and the hall landmark of this disease, visual disturbance. One of the most deleterious effect of IIH is through its effect on optic nerve (papilledema) leading to visual field defect, horizontal double vision and finally decrease of visual acuity. Despite this, these presentations may not appears collectively and patient can come with one or two of vague symptoms as in IIH without papilledema variant[5]. So IIH needs an accurate, trusted, and rapid tool for diagnosis and follow up. Modified Dandy criteria[6,7] gives an informative description for IIH and a differentiation from other causes of increase intracranial pressure through; Signs and symptoms of increased intracranial pressure, Absence of localizing findings on neurologic examination, Absence of deformity, displacement, or obstruction of the ventricular system except for evidence of increased cerebrospinal fluid pressure (greater than 200 mm water)[8]. Normal neuroimaging except for empty sella turcica, optic nerve sheath with filled out CSF spaces, and smooth-walled non flow-related venous sinus stenosis or collapse should lead to another diagnosis, No other cause of increased intracranial pressure present for CSF opening pressure of 200 to 250 mm water.

The clinical presentation of the disease is heterogeneous and often not correlating with the objective findings such as lumbar puncture opening pressure and papilledema. Currently, it is not possible to predict if a patient will respond to medical treatment, or which patients may develop severe permanent visual loss. Papilledema, the only non-invasive objective measurable treatment response, develops with substantial delay compared to intracranial pressure. Therefore, an objective tool indicating permanent optic nerve damage is sorely needed and will help guide treatment and predicting disease outcome. Biomarkers have this advantage as they allow early predicting optic nerve damage. For that reason CSF biomarkers deserve precise understanding for there rule in IIH which is the aim of our study.

ELIGIBILITY:
Inclusion Criteria:

- 1. All patients with signs and symptoms of increased intracranial pressure (headaches, nausea, vomiting, transient visual obscurations, papilledema).

2. CSF opening pressure >25 cm water with normal CSF composition.

Exclusion Criteria:

* 1. localizing neurologic signs, except for unilateral or bilateral sixth cranial nerve palsy.

  2. Evidence of hydrocephalus, mass, infection, structural, or vascular lesion (including venous sinus thrombosis) on imaging.

  3. Patients with IIH who undergo surgical intervention (thecoperitoneal shunt or optic nerve fenestration) 4. Other identified causes of increased ICP.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-11-20 (Actual); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Relation between lumper puncture opening pressure and specific biomarkers | Baseline
  Lumper puncture and measurement of CSF opening pressure (above 20 mm water).
  Measurement tools:
  Enzyme-linked immunosorbent assay (ELISA) test for amount of specific biomarkers both in CSF and serum.
  Specific Biomarkers:
  1. Neurofilament light chain(NLC)
  2. Hypoxia induced factor(HIF)
Relation between lumper puncture opening pressure and visual disturbance | 3 days
  Clinical and visual assessment and CSF opening pressure measurement. measurement tools: Ophthalmoscope Measuring grades of papilledema using the Frisén scale

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud H Ragab, professor, Study Chair — professor; Abdelhakeem A Essa, Ass. prof., Study Director — Assistant professor
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Kalyvas A, Neromyliotis E, Koutsarnakis C, Komaitis S, Drosos E, Skandalakis GP, Pantazi M, Gobin YP, Stranjalis G, Patsalides A. A systematic review of surgical treatments of idiopathic intracranial hypertension (IIH). Neurosurg Rev. 2021 Apr;44(2):773-792. doi: 10.1007/s10143-020-01288-1. Epub 2020 Apr 25. PMID 32335853
- [Background] Sinclair AJ, Ball AK, Burdon MA, Clarke CE, Stewart PM, Curnow SJ, Rauz S. Exploring the pathogenesis of IIH: an inflammatory perspective. J Neuroimmunol. 2008 Sep 15;201-202:212-20. doi: 10.1016/j.jneuroim.2008.06.029. Epub 2008 Aug 3. PMID 18676028